CLINICAL TRIAL: NCT01974752
Title: A Randomised, Double-Blind Study to Assess the Efficacy of Selumetinib (AZD6244: ARRY-142886) (Hyd-Sulfate) in Combination With Dacarbazine Compared With Placebo in Combination With Dacarbazine as First Systemic Therapy in Patients With Metastatic Uveal Melanoma (SUMIT)
Brief Title: Selumetinib (AZD6244: ARRY-142886) (Hyd-Sulfate) in Metastatic Uveal Melanoma (SUMIT)
Acronym: SUMIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1344C00001
Record Dates: First submitted 2013-10-10; First posted 2013-11-04 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic; Uveal Melanoma
Keywords: uveal melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Uveal Melanoma | interventions — AZD 6244; Dacarbazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- selumetinib 75mg twice daily (Experimental): selumetinib 75mg twice daily in combination with dacarbazine.
  Interventions: Drug: 75mg selumetinib; Drug: Dacarbazine
- placebo twice daily (Placebo Comparator): placebo twice daily in combination with dacarbazine.
  Interventions: Drug: placebo; Drug: Dacarbazine

INTERVENTIONS:
Drug: 75mg selumetinib — selumetinib tablets p.o. twice daily taken in combination with dacarbazine 1000mg/m2 iv on day 1 of every 21-day cycle.
  Arms: selumetinib 75mg twice daily
Drug: placebo — placebo tablets p.o. twice daily taken in combination with dacarbazine 1000mg/m2 iv on day 1 of every 21-day cycle.
  Arms: placebo twice daily
Drug: Dacarbazine — dacarbazine 1000mg/m2 iv on day 1 of every 21-day cycle taken in combination with either selumetinib or placebo tablets p.o. twice daily.

SUMMARY:
Selumetinib therapy in patients with metastatic uveal melanoma.

DETAILED DESCRIPTION:
A randomised double-blind study to assess the efficacy of selumetinib (AZD6244, Hyd-Sulfate) in combination with Dacarbazine compared with placebo in combination with Dacarbazine as first systemic therapy in patients with metastatic uveal melanoma (SUMIT)

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of metastatic uveal melanoma; Written consent from female or male patients aged 18 years and over. Histological or cytological confirmation of melanoma who are suitable for treatment with dacarbazine chemotherapy.

* At least one lesion that can be accurately measured at baseline as>/=10mm in the longest diameter. (except lymph nodes which must have short axis ≥15 mm) with CT or MRI and which is suitable for accurate repeated measurements
* ECOG performance status 0-1
* life expectancy >12 weeks
* Normal organ and marrow function
* Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients
* Patients should be able to swallow selumetinib/placebo capsules

Exclusion Criteria:-Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)

* Previous randomisation in the present study
* Patients cannot have previously been treated with a systemic anti-cancer therapy. Patients can have prior intra-hepatic or non-systemic therapy. -Having received any of the following within the specified timeframe:

Any prior systemic anti-cancer therapy for the treatment of this current diagnosis, An investigational drug within 30 days of starting treatment or within five half-lives of the compound (whichever is the most appropriate is at the discretion of the Investigator), or have not recovered from side effects of an investigational drug Any non-systemic anti-cancer therapy which has not been cleared from the body by the time of starting study treatment Radiation therapy within 4 weeks prior to starting study treatment, or limited field of radiation for palliation within 7 days of the first dose of study treatment Major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) which would prevent administration of study treatment, Any prior investigational therapy comprising inhibitors of RAS, RAF or MEK at any time, Previous treatment with dacarbazine. Any unresolved toxicity >CTCAE grade 2 from previous anti-cancer therapy, excluding alopecia -History of allergic reactions attributed to compounds of similar chemical or biologic composition to selumetinib or dacarbazine

--Symptomatic brain metastases or spinal cord compression (patients must be treated and stable off steroids and anti-convulsants for at least 1 month prior to entry into the study)

Cardiac conditions as follows:

* Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy)
* Acute coronary syndrome within 6 months prior to starting treatment
* Uncontrolled Angina - Canadian Cardiovascular Society grade II-IV despite medical therapy - Symptomatic heart failure (New York Heart Association [NYHA] Class II-IV,- Prior or current cardiomyopathy
* Baseline LVEF <55% measured by echocardiography or MUGA. Appropriate correction to be used if a MUGA is performed
* Severe valvular heart disease
* Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
* QTcF >450 ms or other factors that increase the risk of QTc prolongation
* Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* Refractory nausea and vomiting, chronic gastrointestinal diseases (eg inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption
* History of another primary malignancy within 5 years prior to starting study treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study
* Ophthalmologic conditions:
* Current or past history of central serous retinopathy
* Current or past history of retinal vein occlusion
* IOP >21 mmHg or uncontrolled glaucoma (irrespective of IOP)
* Female patients who are breast-feeding a child and male or female patients of reproductive potential who are not employing an effective method of birth control
* Clinical judgement by the Investigator that the patient should not participate in the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Lutherville, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
- Belgium (4):
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Hus, Finland
- France (2):
  - Research Site, Nice
  - Research Site, Paris
- Germany (2):
  - Research Site, Heidelberg
  - Research Site, München
- Israel (2):
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
- Research Site, Leiden, Netherlands
- Spain (4):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Northwood
  - Research Site, Nottingham
  - Research Site, Swansea

REFERENCES:
- [Derived] Carvajal RD, Piperno-Neumann S, Kapiteijn E, Chapman PB, Frank S, Joshua AM, Piulats JM, Wolter P, Cocquyt V, Chmielowski B, Evans TRJ, Gastaud L, Linette G, Berking C, Schachter J, Rodrigues MJ, Shoushtari AN, Clemett D, Ghiorghiu D, Mariani G, Spratt S, Lovick S, Barker P, Kilgour E, Lai Z, Schwartz GK, Nathan P. Selumetinib in Combination With Dacarbazine in Patients With Metastatic Uveal Melanoma: A Phase III, Multicenter, Randomized Trial (SUMIT). J Clin Oncol. 2018 Apr 20;36(12):1232-1239. doi: 10.1200/JCO.2017.74.1090. Epub 2018 Mar 12. PMID 29528792
- [Derived] Carvajal RD, Schwartz GK, Mann H, Smith I, Nathan PD. Study design and rationale for a randomised, placebo-controlled, double-blind study to assess the efficacy of selumetinib (AZD6244; ARRY-142886) in combination with dacarbazine in patients with metastatic uveal melanoma (SUMIT). BMC Cancer. 2015 Jun 10;15:467. doi: 10.1186/s12885-015-1470-z. PMID 26059332

RESULTS

PARTICIPANT FLOW:
Groups:
- Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2: Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2
- Placebo + Dacarbazine 1000 mg/m2: Placebo + Dacarbazine 1000 mg/m2
Period: Overall Study
Arm/Group | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 | Placebo + Dacarbazine 1000 mg/m2
Started | 97 | 32
Completed | 60 | 17
Not Completed | 37 | 15
Not completed — Death | 33 | 11
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Other Eligibility Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 | Placebo + Dacarbazine 1000 mg/m2 | Total
Number analyzed (Participants) | 97 | 32 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (12.28) [42 to 84] | 59.6 (11.28) [22 to 86] | 60.6 (12.01) [22 to 86]
Age, Customized [Number; unit: Participants]
  <55 years | 26 | 11 | 37
  >=55 years To <65 years | 25 | 9 | 34
  >=65 years | 46 | 12 | 58
Gender [Count of Participants; unit: Participants]
  Female | 42 | 19 | 61
  Male | 55 | 13 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  Other | 1 | 1 | 2
  White | 96 | 31 | 127

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Efficacy of Selumetinib in Combination With Dacarbazine Compared With Placebo in Combination With Dacarbazine Measured as Progression Free Survival (PFS) Using BICR According to RECIST 1.1.
Description: Progression free survival (PFS) using blinded independent central review (BICR) according to the Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1). Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From Randomization, then every 6 weeks up until progression or death (whichever is sooner) assessed up to 15th May 2015
Population: All randomised patients and will compare the treatment groups on the basis of randomised treatment, regardless of the treatment actually received. Note, this is also known as the Full Analysis set (FAS).
Measure: Number; unit: number of progression events
Arm/Group | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 | Placebo + Dacarbazine 1000 mg/m2
Number analyzed (Participants) | 97 | 32
number of progression events | 82 [2.8 to 2.8] | 24 [1.8 to 1.8]
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 vs Placebo + Dacarbazine 1000 mg/m2; Test type: Superiority or Other; p = 0.3195, Log Rank; Factor for treatment and liver metastases; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.48 to 1.27] — A hazard ratio < 1 favours Selumetinib in combination with Dacarbazine

2. Secondary Outcome: Assessment of the Efficacy of Selumetinib in Combination With Dacarbazine Compared With Placebo in Combination With Dacarbazine in Terms of Objective Response Rate (ORR) by BICR
Description: ORR at Week 6 using BICR according to RECIST 1.1
Time Frame: From Randomization, then every 6 weeks up until progression or death (whichever is sooner) assessed up to 15th May 2015
Population: Full Analysis Set
Measure: Number; unit: number of responders
Arm/Group | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 | Placebo + Dacarbazine 1000 mg/m2
Number analyzed (Participants) | 97 | 32
number of responders | 3 | 0

3. Secondary Outcome: Assessment of the Efficacy of Selumetinib in Combination With Dacarbazine Compared With Placebo in Combination With Dacarbazine in Terms of Change in Tumour Size at Week 6 by BICR
Description: Percent change in tumour size at Week 6 using BICR according to RECIST 1.1
Time Frame: From Randomization, then every 6 weeks up until progression or death (whichever is sooner) assessed up to 15th May 2015
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 | Placebo + Dacarbazine 1000 mg/m2
Number analyzed (Participants) | 92 | 27
percent change | 6.94 (18.001) [6.94 to 6.94] | 19.76 (38.264) [19.76 to 19.76]
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 vs Placebo + Dacarbazine 1000 mg/m2; Test type: Superiority or Other; p = 0.1284, ANCOVA; ANCOVA of log (W6/BL) tumour assessments with a factor for trt, and covariates for liver mets, log BL tumour size, and time from BL scan to rand; Geometric LS mean ratio = 0.94, 95% CI 2-sided [0.88 to 1.02] — A geometric least squares mean ratio < 1 favours Selumetinib in combination with Dacarbazine

4. Secondary Outcome: Assessment of the Overall Survival (OS) in Patients Taking Selumetinib in Combination With Dacarbazine Compared With Those Taking Placebo in Combination With Dacarbazine
Description: Overall Survival
Time Frame: From Randomization, up until death assessed up to 15th May 2015
Population: as for outcome 1
Measure: Number; unit: Number of Overall Survival Events
Arm/Group | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 | Placebo + Dacarbazine 1000 mg/m2
Number analyzed (Participants) | 97 | 32
Number of Overall Survival Events | 34 | 14
Statistical Analysis 1: Comparison: Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 vs Placebo + Dacarbazine 1000 mg/m2; Test type: Superiority or Other; p = 0.4011, Log Rank; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.39 to 1.46]

ADVERSE EVENTS:
Time Frame: From informed consent up until end of double blind period
Arm/Group | Placebo + Dacarbazine 1000 mg/m2 | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2
Serious Adverse Events (participants affected / at risk) | 2/32 | 20/97
Other Adverse Events (participants affected / at risk) | 32/32 | 97/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Dacarbazine 1000 mg/m2 (N=32) | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 (N=97)
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 2 (2)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Dacarbazine 1000 mg/m2 (N=32) | Selumetinib 75 mg BD + Dacarbazine 1000 mg/m2 (N=97)
ANAEMIA (Blood and lymphatic system disorders) | 4 (6) | 18 (22)
NEUTROPENIA (Blood and lymphatic system disorders) | 11 (14) | 25 (35)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 26 (39)
CONSTIPATION (Gastrointestinal disorders) | 14 (19) | 37 (46)
ASTHENIA (General disorders) | 4 (5) | 20 (21)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 (3) | 6 (6)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (4) | 4 (5)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
PARAESTHESIA (Nervous system disorders) | 2 (4) | 5 (5)
INSOMNIA (Psychiatric disorders) | 4 (4) | 8 (8)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 19 (23)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (12)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
VISION BLURRED (Eye disorders) | 1 (1) | 10 (11)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 11 (12)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (4) | 8 (8)
DIARRHOEA (Gastrointestinal disorders) | 7 (11) | 43 (83)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 9 (9)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 11 (12)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 5 (5)
NAUSEA (Gastrointestinal disorders) | 6 (12) | 60 (92)
STOMATITIS (Gastrointestinal disorders) | 2 (2) | 15 (16)
VOMITING (Gastrointestinal disorders) | 6 (7) | 27 (36)
CHILLS (General disorders) | 1 (1) | 5 (6)
FACE OEDEMA (General disorders) | 0 (0) | 6 (7)
FATIGUE (General disorders) | 15 (16) | 43 (49)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 42 (47)
PYREXIA (General disorders) | 5 (6) | 8 (9)
HEPATIC PAIN (Hepatobiliary disorders) | 3 (3) | 3 (3)
BRONCHITIS (Infections and infestations) | 0 (0) | 5 (5)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 5 (6)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 9 (9)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (7) | 28 (36)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 5 (8) | 29 (36)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (3) | 8 (8)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 36 (40)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 6 (8)
PLATELET COUNT DECREASED (Investigations) | 3 (4) | 7 (10)
WEIGHT DECREASED (Investigations) | 2 (2) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 (9) | 17 (18)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (3) | 5 (6)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (2) | 6 (8)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 5 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (10)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 12 (14)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3)
DIZZINESS (Nervous system disorders) | 3 (3) | 6 (7)
DYSGEUSIA (Nervous system disorders) | 3 (4) | 11 (11)
HEADACHE (Nervous system disorders) | 3 (3) | 13 (13)
SYNCOPE (Nervous system disorders) | 0 (0) | 6 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 9 (9)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 30 (37)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (5) | 14 (15)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 55 (60)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (14)
HYPERTENSION (Vascular disorders) | 2 (2) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No